CLINICAL TRIAL: NCT05331781
Title: Comparative Study Between Ultrasound-Guided Transversus Abdominis Plane Block and Spinal Morphine for Pain Relief After Elective Caesarean Section
Brief Title: Ultrasound-Guided TAP Block and Spinal Morphine for Pain Relief After Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Mokhtar Ahmed, lecturer of anesthesia and intensive care, Sohag University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: soh-Med-22-2-41
Record Dates: First submitted 2022-04-02; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Post Operative Pain
Keywords: Ultrasound-Guided Transversus Abdominis Plane Block, Morphine, Caesarean section
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversus abdominis plain block group (Experimental): post-cesarean section tap block will be given by ultrasound guidance using 20 ml bupivacaine local anesthetic 0.25% concentration for each side as an adjuvant to spinal anesthesia
  Interventions: Procedure: Ultrasound-Guided Transversus Abdominis Plane Block
- intrathecal morphia group (Experimental): intrathecal 150 microgram morphine in a 0.5 ml volume as an adjuvant to spinal anesthesia
  Interventions: Drug: Morphine

INTERVENTIONS:
Procedure: Ultrasound-Guided Transversus Abdominis Plane Block — patient in the supine position, ultrasound will be used to identify the plane between the internal oblique and transversus abdominis muscle to inject 20 ml of local anesthetic for each side
  Arms: transversus abdominis plain block group
Drug: Morphine — intrathecal 150 microgram morphine in a 0.5 ml volume will be added to bupivacaine as an adjuvant to spinal anesthesia
  Arms: intrathecal morphia group

SUMMARY:
This interventional double-blind randomized controlled study was carried out on 60 cases underwent elective caesarean section delivery, they were divided into 2 groups; patients were randomly allocated into two equal groups; Group M: received intrathecal 150 microgram morphine in a 0.5 ml volume, mixed with 10 mg of hyperbaric bupivacaine 0.5 % in a 2 ml volume (total volume 2.5 ml). Group B: received intrathecal 10 mg hyperbaric bupivacaine 0.5% 2ml volume + 0.5 saline (Total volume 3ml) and at the end of surgery patient received bilateral TAP block with 20 ml volume of 0.25% bupivacaine on each side.

ELIGIBILITY:
Inclusion Criteria:

* pregnant females scheduled for elective cesarean section

Exclusion Criteria:

* Patient refusal Patients with known allergies or with past history of allergy to local anesthesia Patients having an infection at the site of injection either in the back or in the abdominal region, Patients with coagulopathy or on systemic anticoagulation, Chronic opioid abuse, significant neurological, psychiatric or neuromuscular disease, Drug abuse and alcoholism, Obesity (BMI 30 and higher), Cardiovascular disease and Endocrine disorders.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
prevention of post-operative pain | 72 hours
  reduction of visual analogue scale post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No